CLINICAL TRIAL: NCT06062836
Title: The Platform for Interdisciplinary Cardiovascular-metabolic-neurovascular Diseases (PICMAN) Across National University Health System (NUHS)
Brief Title: The Platform for Interdisciplinary Cardiovascular-metabolic-neurovascular Diseases (PICMAN)
Acronym: PICMAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: PICMAN
Record Dates: First submitted 2023-04-10; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-04

CONDITIONS: Cardiometabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Molecular phenotyping via
  1. Analysis of peripheral blood mononuclear cells (PBMC) for immunometabolic profile analysis
  2. Analysis of genomics and microbiome analysis using exosome isolates, stool and urine samples
  3. "Omits" profiling covering their genomics, epigenomics, transcriptomics, and proteomics via differentiation of patient-derived iPSCs into cardiac cell-types
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Changes in metabolism and mitochondrial function appear to precede cardiac dysfunction, with much evidence supporting metabolic dysregulation as one of the earliest precursors of cardiovascular disease. We hypothesise that quantifiable metabolic inflexibility may be representative of an individual in his/her silent, but high-risk progression towards insulin resistance, diabetes and cardiovascular disease. The platform for interdisciplinary cardiovascular-metabolic-neurovascular diseases (PICMAN) across National University Health System (NUHS) is a pilot, prospective, multi-ethnic cohort study in Singapore.

Through extensive phenotyping in a preventive cardiology cohort, the central aim is to define the metabolic flexibility range in a cohort of individuals at elevated risk of atherosclerotic cardiovascular disease, to correlate metabolic flexibility to measures of cardiometabolic health, including diastolic dysfunction, coronary and cerebral atherosclerosis, body fat distribution and severity of non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Aims

1. Define norms for metabolic flexibility in a multi-ethnic Southeast Asian cohort of individuals without manifest ASCVD
2. Understand the association of metabolic inflexibility with cardiovascular measures of diastolic dysfunction and coronary and cerebral atherosclerosis
3. Understand the association of metabolic inflexibility with measures of body fat distribution
4. Understand the correlation between metabolic flexibility and insulin sensitivity along the spectrum of subclinical cardiovascular disease and severity of non-alcoholic fatty liver disease
5. Associations of the gut microbiome as well as metabolomic and molecular markers with cardio-cerebrovascular measures, metabolic flexibility and liver fibrosis

The PICMAN study seeks to lay the foundations for further future larger scale and more experimentally ambitious studies based on the overarching hypothesis that metabolic flexibility is an early marker in subclinical cardiovascular disease, indicating a point of timely intervention where the disease process is still reversible. The importance of a deeply-phenotyped local cohort will allow us to study the progression of CVD in seemingly well adults, converging imaging, biochemical, metabolic markers, and 'omics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-70 at screening
* 10-year ASCVD risk > 5% measured by QRISK 3 calculator

Exclusion Criteria:

* Established DM (Prior diagnosis, long term medications or HbA1c >=6.5)
* Established CVD, such as ischemic heart disease, cerebrovascular accident, heart failure, atrial fibrillation
* Pregnancy
* Known contraindications to CT scan, such as allergy to contrast

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants between the ages of 21 and 70 at screening without a prior history of MACE, coronary artery disease diagnosis, established diabetes, with a calculated 10-year ASCVD risk > 5% based on QRISK3 calculator are eligible for PICMAN. Recruitment of individuals takes place at NUHS, where community-dwelling individuals without cardiac disease will be referred via outreach to primary care and community partners in Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Metabolic flexibility | Up to 5 years
  Metabolic flexibility will be calculated (deltaRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Mayank Dalakoti, Principal Investigator — National University Health System; Roger Foo, Principal Investigator — National University Health System
Locations (1):
- National University Health System, Singapore, Singapore